CLINICAL TRIAL: NCT01060683
Title: Liver Resection and Non-invasive Measurement of Hemoglobin Concentration With Pulse Co-oximetry
Brief Title: Non-invasive Measurement of Hemoglobin Concentration With Pulse Co-oximetry
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: SpHb-001
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Elective Hepatic Resection
Keywords: hemoglobin; Coagulation variables; blood chemistry; Blood gas analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — laboratory hemoglobin, Coagulation variables,blood chemistry,Blood gas analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: 15 patients: for elective hepatic resection
  Interventions: Biological: Hemoglobin determination + NaCl 0.9% bolus
- Group 2: 15: for elective hepatic resection
  Interventions: Biological: hemoglobin determination + Venofundin bolus

INTERVENTIONS:
Biological: Hemoglobin determination + NaCl 0.9% bolus
  Groups: Group 1: 15 patients
Biological: hemoglobin determination + Venofundin bolus
  Groups: Group 2: 15

SUMMARY:
The purpose of this study is to evaluate the accuracy of continuous SpHb measurement ( Rainbow DCI, Masimo, Irvine Ca, USA) compared to the current method of monitoring (blood sampling), both during phases of hemoconcentration and hemodilution.

ELIGIBILITY:
Inclusion Criteria:

* All patients: Age > 18 years
* ASA class I and II patient requiring hepatic resection

Exclusion Criteria:

* Patient refusal
* Patients with a perioperative blood loss exceeding 5ml/kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA class I and II patients for elective hepatic resection
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the accuracy of continuous SpHb measurement during hepatic resection compared with standard (invasive) Hb measurement | during operation

SECONDARY OUTCOMES:
the effect of a bolus of crystalloid on SpHb level will be compared to the effect of a bolus of colloid on the SpHb level. | during operation

CONTACTS AND LOCATIONS:
Overall Officials: Herman G.D. Hendriks, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen,University of Groningen, the Netherlands, Groningen, Netherlands

REFERENCES:
- [Derived] Vos JJ, Kalmar AF, Struys MM, Wietasch JK, Hendriks HG, Scheeren TW. Comparison of arterial pressure and plethysmographic waveform-based dynamic preload variables in assessing fluid responsiveness and dynamic arterial tone in patients undergoing major hepatic resection. Br J Anaesth. 2013 Jun;110(6):940-6. doi: 10.1093/bja/aes508. Epub 2013 Jan 24. PMID 23348202